CLINICAL TRIAL: NCT03000270
Title: Door To Unloading With IMPELLA CP System in Acute Myocardial Infarction to Reduce Infarct Size (DTU): A Prospective Feasibility Study
Brief Title: Door To Unloading With IMPELLA CP System in Acute Myocardial Infarction - Safety and Feasibility Study
Acronym: DTU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abiomed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DTU - Safety and Feasibility
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2018-11

CONDITIONS: STEMI
Keywords: Infarct Size; Impella; Unloading; Left Ventricle; PPCI; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Prolonged unloading prior to PPCI (Active Comparator): Activation of Impella CP for a 30 minute duration prior to primary percutaneous coronary intervention
  Interventions: Device: Impella unloading prior to PPCI
- Immediate unloading prior to PPCI (Active Comparator): Activation of Impella CP immediately prior to primary percutaneous coronary intervention
  Interventions: Device: Impella unloading prior to PPCI

INTERVENTIONS:
Device: Impella unloading prior to PPCI — Impella unloading prior to PPCI

SUMMARY:
Direct active unloading of the left ventricle with the Impella CP System prior to PPCI in patients with ST-elevation myocardial infarction (STEMI) is safe and feasible

DETAILED DESCRIPTION:
A multi-center, prospective, randomized, two-arm feasibility trial to assess the potential role of unloading with the Impella CP prior to revascularization in reducing infarct size. The study design includes 1:1 randomization between: 1) Delay Arm: 30 minutes of unloading with Impella CP prior to primary percutaneous coronary intervention (PPCI); and 2) Immediate Arm: initiation of Impella CP unloading followed immediately by PPCI.

Study Hypothesis: Direct active unloading of the left ventricle with the Impella CP System prior to PPCI in patients with ST-elevation myocardial infarction (STEMI) is safe and feasible

ELIGIBILITY:
Main Inclusion Criteria:

* Age 21-80 years
* First myocardial infarction
* Acute anterior STEMI with ≥ 2 mm in 2 or more contiguous anterior leads or≥ 4 mm total ST-segment deviation sum in the anterior leads
* Signed Informed Consent

Main Exclusion Criteria:

* Cardiogenic shock defined as: systemic hypotension (systolic BP less than 90 mmHg or the need for inotropes/pressors to maintain a systolic BP Greater than 90mmHg) plus one of the following: any requirement for pressors/inotropes prior to arrival at the cath lab, clinical evidence of end organ hypoperfusion, lactate level greater than 2.5mmol/L
* Inferior STEMI or suspected right ventricular failure
* Suspected or known pregnancy
* Suspected active infection
* History or known hepatic insufficiency prior to catheterization
* On dialysis therapy
* Known contraindication to:
* Undergoing MRI or use of gadolinium
* Heparin, pork, pork products or contrast media
* Receiving a drug-eluting stent
* Participation in the active treatment or follow-up phase of another clinical study of an investigational drug or device

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-06-19 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Infarct size at 30 Days | 30 Days
  Assessment of infarct size as percent of left ventricular (LV) mass, evaluated using CMR, at 30 days post-PPCI
MACCE at 30 Days | 30 Days
  A composite of the following Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) at 30 days:
  * Cardiovascular mortality
  * Re-infarction
  * Stroke/TIA
  * Major vascular complication

SECONDARY OUTCOMES:
Infarct Characteristics - LV mass | 3 - 5 and 30 Days
  Using CMR at 3-5 & 30 days, assessement of Infarct size as a percent of LV mass
Infarct Characteristics - area at risk | 3 - 5 and 30 Days
  Using CMR at 3-5 & 30 days, assessment of Infarct size as a percent of area (myocardium) at risk,
30 Day Safety Endpoint Rates | 30 Days
  Event rate for All-cause mortality, Cardiovascular mortality, Re-infarction, Stroke/TIA, Vascular complications, Worsening heart failure or hemodynamic compromise requiring inotropic or hemodynamic support post Impella explant, Repeat revascularization, Aortic valve injury or dysfunction, Renal failure, Hemolysis, Hematoma, Bleeding, Thrombocytopenia
Infarct Characteristics microvascular obstruction | 3-5 and 30 Days
  Using CMR at 3-5 & 30 days, measurement of percent of microvascular obstruction (%MVO)
Left Ventricular Function- LV end systolic and diastolic volume index | 3-5 and 30 Days
  Using CMR imaging post PCI: assessment of LV end systolic and diastolic volume index (LVESVi & LVEDVi)
Left Ventricular Function - Ejection Fraction | 3-5 and 30 Days
  Using CMR at 3-5 & 30 days post PCI: assessment of Ejection fraction (EF)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - Wellstar/Kennestone Hospital, Marietta, Georgia
  - Detroit Medical Center, Detroit, Illinois
  - Advocate Edward Hospital, Oakbrook Terrace, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - ABIOMED, Inc., Danvers, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Spectrum, Grand Rapids, Michigan
  - Hackensack Medical Center, Hackensack, New Jersey
  - University of Buffalo Hospital, Buffalo, New York
  - Northwell Health, Manhasset, New York
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kapur NK, Alkhouli MA, DeMartini TJ, Faraz H, George ZH, Goodwin MJ, Hernandez-Montfort JA, Iyer VS, Josephy N, Kalra S, Kaki A, Karas RH, Kimmelstiel CD, Koenig GC, Lau E, Lotun K, Madder RD, Mannino SF, Meraj PM, Moreland JA, Moses JW, Kim RL, Schreiber TL, Udelson JE, Witzke C, Wohns DHW, O'Neill WW. Unloading the Left Ventricle Before Reperfusion in Patients With Anterior ST-Segment-Elevation Myocardial Infarction. Circulation. 2019 Jan 15;139(3):337-346. doi: 10.1161/CIRCULATIONAHA.118.038269. PMID 30586728
- See also: Unloading the Left Ventricle Before Reperfusion in Patients With Anterior ST-Segment-Elevation Myocardial Infarction. — http://www.ahajournals.org/doi/10.1161/CIRCULATIONAHA.118.038269